CLINICAL TRIAL: NCT07201116
Title: Effectiveness of a Geographic Information System-Integrated Mobile Platform for Coordinating Early Stage Rehabilitation After Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Health-GIS Platform for Hip Replacement Rehabilitation Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulip Medicine (Other)
Responsible Party: Principal Investigator, Didar Khassenov, Head of department, Tulip Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: NROC 4
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Hip Arthroplasty Replacement; Hip Arthroplasty, Total; Rehabilitation; Hip Osteoarthritis
Keywords: Total hip arthroplasty; Hip replacement; Rehabilitation; Patient navigation; Mobile health application; Geographic information systems; Healthcare delivery; Rehabilitation access; Post-operative care; Quality of life
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GIS-Guided Rehabilitation App (Experimental): Patients receive access to a specialized mobile application with integrated Geographic Information System (GIS) components for rehabilitation service coordination after total hip arthroplasty.
  Interventions: Device: Health-GIS Rehabilitation Coordination Platform
- Standard Primary Care Referral (Active Comparator): Patients receive standard rehabilitation referral process through primary care physicians after total hip arthroplasty
  Interventions: Other: Standard Rehabilitation Referral

INTERVENTIONS:
Device: Health-GIS Rehabilitation Coordination Platform — Participants receive access to a specialized mobile application with integrated Geographic Information System (GIS) components for rehabilitation service coordination. While hospitalized, patients submit rehabilitation requests through the platform, indicating their location, desired time, and specific rehabilitation needs. Registered rehabilitation centers within the platform receive these requests and can submit counter-proposals with available slots, services offered, and estimated costs. The platform provides real-time visualization of available rehabilitation facilities on an interactive map, displays facility ratings, services offered, current capacity, and waiting times. Patients receive automated notifications about new proposals and can compare options based on location proximity, service quality ratings, and availability. Technical support is available through in-app messaging and a dedicated helpline during business hours.
  Arms: GIS-Guided Rehabilitation App
Other: Standard Rehabilitation Referral — Upon discharge, patients receive written recommendations stating that rehabilitation is advised as part of their post-operative care plan. No specific rehabilitation facilities are recommended or contacts provided by the surgical team. Patients are instructed to contact their assigned primary care physician (general practitioner) at their local polyclinic for further referral coordination. The primary care physician is responsible for identifying available rehabilitation facilities, making referrals, and coordinating the rehabilitation timeline based on their knowledge of local resources and current availability. This intervention represents routine clinical practice typically provided to patients after total hip arthroplasty.
  Arms: Standard Primary Care Referral

SUMMARY:
This study tests whether a mobile phone app with mapping technology can help patients find rehabilitation services faster after hip replacement surgery. After having their hip replaced, patients typically need several months of physical therapy to recover fully. However, many patients face long waiting times or don't know where to find rehabilitation services near them.

In this study, half of the patients will use a new mobile app that shows rehabilitation centers on a map, displays available appointment times, and allows patients to compare services and costs. The other half will receive standard care, where they must contact their family doctor to help find rehabilitation services.

The study will measure how quickly patients start rehabilitation after leaving the hospital, how well their hip functions after treatment, their quality of life, and pain levels. The investigators will also look at whether the app is easy to use.

DETAILED DESCRIPTION:
Total hip arthroplasty (hip replacement) is one of the most successful surgical procedures in modern orthopedics, with over 528 million people worldwide affected by osteoarthritis requiring joint replacement. The demand is projected to increase dramatically: 71% growth in the US by 2030 (635,000 procedures), 198% growth in Australia by 2046 (94,086 procedures), and 99-147% growth in Japan by 2030 depending on demographic groups.

Success of hip replacement surgery largely depends on timely access to rehabilitation services, particularly during the early recovery period (first 3-6 months post-surgery). Current medical rehabilitation principles emphasize early initiation, continuity, and seamless care coordination to optimize clinical outcomes. However, healthcare systems worldwide face significant challenges in organizing effective rehabilitation services.

The primary objective is to evaluate the effectiveness of implementing a GIS-integrated rehabilitation coordination platform for organizing early-stage rehabilitation after total hip arthroplasty. The investigators hypothesize that using a specialized mobile application with integrated GIS components will eliminate information gaps, ensure equitable patient flow distribution among medical organizations, reduce time from surgical discharge to second-stage rehabilitation initiation, and consequently improve functional treatment outcomes while enhancing healthcare system resource utilization efficiency.

After discharge from surgical hospitals, patients often encounter an information vacuum regarding available rehabilitation services. Primary care physicians typically have limited knowledge of regional rehabilitation centers, severely restricting patient routing options. This leads to systematic violations of key rehabilitation principles - early initiation and continuity of care - negatively impacting surgical outcomes.

Kazakhstan's healthcare system exemplifies these challenges, with critical imbalances between rehabilitation service demand and supply. Leading national centers performing thousands of hip replacements annually can provide rehabilitation to only a small fraction of patients, creating waiting lists extending several months. This disproportion generates systematic risks and healthcare delivery violations, with over 5.9 million healthcare delivery defects identified in 2024, including inappropriate service volume increases, unjustified medical care provision, and deviations from clinical protocols.

Healthcare digitalization offers innovative solutions to these systemic problems. Geographic Information Systems (GIS) have been successfully applied in various medical fields for analyzing spatial distribution of medical resources, optimizing patient routing, and improving service accessibility. A rehabilitation coordination platform with integrated GIS components could fundamentally transform rehabilitation service organization by providing transparency regarding available services, real facility capacity, and care accessibility.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Completed primary total hip arthroplasty within the past 6 months
* Ability to understand study procedures and provide signed informed consent
* Fluency in Russian or Kazakh language
* Access to smartphone or tablet device with internet connectivity

Exclusion Criteria:

* Severe cognitive impairment
* Participation in another clinical trial that might interfere with study outcomes
* Intraoperative or postoperative complications requiring extended hospitalization after total hip arthroplasty
* Medical contraindications to rehabilitation
* Planned total hip arthroplasty within 12 months
* Severe visual impairments preventing mobile application usage
* Patients who declined to participate after being informed about the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Time to Rehabilitation Initiation | 12 months from enrollment
  Time from discharge from surgical hospital to initiation of second-stage rehabilitation services, measured in days
SF-12 Quality of Life Score | Baseline, 6 months, and 12 months from enrollment
  12-Item Short Form Health Survey (SF-12) Physical Component Summary (PCS): 0-100 Mental Component Summary (MCS): 0-100 Higher scores indicate better quality of life and better health status.

SECONDARY OUTCOMES:
Harris Hip Score | Baseline, 6 weeks, 6 months, and 12 months from enrollment
  Functional outcome assessment measuring hip joint function, pain, and mobility. The scale ranges from 0 to 100, with higher scores indicating better hip function and less disability.
Visual Analog Scale (VAS) Pain Score | Baseline, 6 weeks, 6 months, and 12 months from enrollment
  Pain intensity assessment using a 0-10 scale where 0 represents no pain and 10 represents maximum possible pain.
System Usability Scale (SUS) Score | 3 months and 6 months from enrollment
  Usability assessment of the Health-GIS platform for both patients and healthcare facilities. The scale ranges from 0 to 100, with higher scores indicating better usability and user satisfaction.
Quality-Adjusted Life Years (QALY) | 12 months from enrollment
  Health utility measured using SF-6D utility scores derived from SF-12 questionnaire, calculated using the area under the curve method over the 12-month study period The QALY score will range from 0 to 1. A higher QALY score represents a better overall health outcome over the 12-month period, indicating more time spent in a better state of health.

CONTACTS AND LOCATIONS:
Locations (1):
- NCJSC "Astana Medical University", Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No